CLINICAL TRIAL: NCT03597724
Title: Identification of Critical Outcomes in Sarcopenia: a Discrete Choice Experiment
Brief Title: Identification of Critical Outcomes in Sarcopenia
Acronym: DCE-Sarcopenia
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0080; 2018-A00530-55 (Other: ID-RCB)
Record Dates: First submitted 2018-07-10; First posted 2018-07-24 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient suffering from sarcopenia: Subjects aged 65 years or older suffering from sarcopenia (diagnosis performed with a valid definition and valid cut-off points) and they will respond to the Questionnaire composed of 13 choice questions.
  Interventions: Other: Questionnaire composed of 13 choice questions.

INTERVENTIONS:
Other: Questionnaire composed of 13 choice questions. — In this Discrete Choice Experiment (DCE), patients will be asked to choose which one of two hypothetical patients (Patient A and Patient B) suffering from sarcopenia with different levels of outcomes deserves the most the treatment. After completion of the choice tasks, respondents will be asked how difficult they found the choice tasks on a seven-point scale and to questions on their socio-economic and disease characteristics.

SUMMARY:
Patients will be recruited on each site according to inclusion criteria. Participants willing to participate will received an information sheet and a consent form. After given their consent to participate, they will receive a questionnaire composed of 13 choice questions. In this DCE, patients will be asked to choose which one of two hypothetical patients (Patient A and Patient B) suffering from sarcopenia with different levels of outcomes deserves the most the treatment. After completion of the choice tasks, respondents will be asked how difficult they found the choice tasks on a seven-point scale and to questions on their socio-economic and disease characteristics.

DETAILED DESCRIPTION:
The participants will first receive an information letter and consent form. Participants will be free to ask any questions to the doctor/researcher. Once the consent form signed, participants will receive the questionnaire and will be asked to complete it. Explanation of the task and an example choice task should be provided by a doctor or a researcher but the questionnaire is intended to be self-administered. Nevertheless, some level of support can be brought if necessary.

The questionnaire is composed by a general explanation of the purpose of the study followed by a definition of sarcopenia and a clear description of the DCE task. The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided. Each patient will then receive 13 choice sets. After completion of the choice tasks, respondents will be asked how difficult they found the choice tasks on a seven-point scale. Participants who graded the level of difficulty as "extremely difficult" will be removed from the analyses. The DCE task is presented in Appendix 1. The questionnaire also asks questions on patients' characteristics.

The questionnaire has been created with experts during the phase of "Identification and prioritization of important outcomes of sarcopenia". Five attributes and different levels of consequences have been identified by the panel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diagnosis of sarcopenia :
* Muscle mass
* Muscle strength and physical performance should be measured

Exclusion Criteria:

* Problem of Cognitive function
* Diagnosis of dementia
* unability to understand the study and the the questionnaire
* unability to fill in the questionnaire
* major depression

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Population suffering from diagnosed sarcopenia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Quality of life of the patient who are living with Sarcopenia | 1 hour
  Good, Fair, Poor : the choices in the questionnaire The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided The quality of life is one of the five attributes and different levels of consequences have been identified by the panel.

SECONDARY OUTCOMES:
Mobility | 1 hour
  The questionnaire is composed by a general explanation of the purpose of the study followed by a definition of sarcopenia and a clear description of the DCE task. The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided. Each patient will then receive 13 choice sets. After completion of the choice tasks, respondents will be asked how difficult they found the choice tasks on a seven-point scale Possibilities in the questionnaire for the mobility part : Outdoor without difficulties, Outdoor with difficulties, Indoor only, Chairbound, Bedbound The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided The mobility is one of the five attributes and different levels of consequences have been identified by the panel.
Capacity of doing domestic activities | 1 hour
  The questionnaire is composed by a general explanation of the purpose of the study followed by a definition of sarcopenia and a clear description of the DCE task. The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided. Each patient will then receive 13 choice sets. After completion of the choice tasks, respondents will be asked how difficult they found the choice tasks on a seven-point scale Possibilities in the questionnaire for the capacity of doing domestic activities: Manage without difficulties, Manage with difficulty, Unable for domestic activities such as cooking, cleaning, gardening The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided The capacity of doing domestic activities is one of the five attributes and different levels of consequences have been identified by the panel.
The level of Fatigue | 1 hour
  The questionnaire is composed by a general explanation of the purpose of the study followed by a definition of sarcopenia and a clear description of the DCE task. The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided. Each patient will then receive 13 choice sets. After completion of the choice tasks, respondents will be asked how difficult they found the choice tasks on a seven-point scale.
  In the questionnaire the patient chooses between different options for fatigue when doing activities such as walking : Tired not at all, Moderately tired, Tired very easily The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided The level of fatigue is one of the five attributes and different levels of consequences have been identified by the panel.
Incidence of falls | 1 hour
  The questionnaire is composed by a general explanation of the purpose of the study followed by a definition of sarcopenia and a clear description of the DCE task. The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided. Each patient will then receive 13 choice sets. After completion of the choice tasks, respondents will be asked how difficult they found the choice tasks on a seven-point scale It can be Never, Occasional or Frequent in the questionnaire. The attributes and levels are carefully explained in the introduction part of the questionnaire and an example of a completed choice set is provided The incidence of falls is one of the five attributes and different levels of consequences have been identified by the panel.

CONTACTS AND LOCATIONS:
Overall Officials: Rolland Yves, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No